CLINICAL TRIAL: NCT03761472
Title: Comparison of Hyaluronic Acid and Platelet-rich Plasma Injection on Pain, Physical Function and Femoral Cartilage Thickness in Patients With Osteoarthritis
Brief Title: Comparison of Hyaluronic Acid and Platelet-rich Plasma Injections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 71306642-050.01.04-
Record Dates: First submitted 2018-11-23; First posted 2018-12-03 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Knee Osteoarthritis
Keywords: Osteoarthritis; Hyaluronic acid; Platelet-rich plasma; Injection
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Hyaluronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Hyaluronic acid injection (Active Comparator): Hyaluronic acid 48 mg 2.0% in 2 ml solution, once initially.
  Interventions: Biological: Hyaluronic acid injection
- Platelet-rich plasma injection (Active Comparator): Platelet-rich plasma 5 ml, once initially
  Interventions: Biological: Platelet-rich plasma injection
- Unaffected side Hyaluronic acid (No Intervention): Unaffected sides of the patients will be controls for hyaluronic acid group, no intervention.
- Unaffected side Platelet-rich plasma (No Intervention): Unaffected sides of the patients will be controls for Platelet-rich plasma group, no intervention.

INTERVENTIONS:
Biological: Hyaluronic acid injection — Hyaluronic acid 48 mg 2.0% in 2.4 ml solution
  Other Names: Reviscon Mono
  Arms: Hyaluronic acid injection
Biological: Platelet-rich plasma injection — Platelet-rich plasma injection 5ml
  Arms: Platelet-rich plasma injection

SUMMARY:
This study aims to compare the effects of hyaluronic acid injection and platelet rich plasma injection in terms of pain, physical function and femoral cartilage thickness in short term treatment in patients with knee osteoarthritis.

DETAILED DESCRIPTION:
Platelet-rich plasma and hyaluronic acid injections are both popular treatments and commonly used for treatment of knee osteoarthritis. Even though there are many studies investigating the effectiveness of these treatments, the results are mostly qualitative. Also there are a few studies comparing these two treatment modalities. In this study the investigators aim to compare these modalities both for self-reported data (pain, physical function) and objective measurement data (femoral cartilage thickness via ultrasonography). Patients with unilateral osteoarthritis/unilateral complaint will be included in the study. Unaffected side will be controls for each group.

ELIGIBILITY:
Inclusion Criteria:

* Subject is able to consent
* Subject meets Osteoarthritis Research Society International (OARSI) criteria for knee osteoarthritis
* Subject has radiographic Kellgren-Lawrence grade 2-3 osteoarthritis
* Unilateral osteoarthritis/complaint

Exclusion Criteria:

* Past or actual knee infection
* History of surgery, fracture on knee
* Collagen tissue disease
* Systemic inflammatory disease (rheumatoid arthritis, spondyloarthritis etc.)
* Systemic diseases (diabetes, hematologic diseases, endocrinopathies, renal failure, liver failure)
* Knee injection in past 6 months
* Immunodeficiency
* Pregnant/breastfeeding
* Malignancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-01-13 (Actual); Study Completion 2020-01-13 (Actual)

PRIMARY OUTCOMES:
Change of numeric rating scale (rest, movement) | 0, 1st, 6th, months
  Self reported pain scored between 0 (minimum)-10 (maximum). Higher scores represent a worse outcome.
Change of Western Ontario and McMaster Universities Osteoarthritis Index score(WOMAC) | 0, 1st, 6th months
  Self reported questionnaire investigating 24 daily living activities. Each item is scored 0-5 (0:none 5:worst). Yielding a total between 0-100. Higher scores represent a worse outcome.
Change of femoral cartilage thickness via ultrasonography. | 0, 1st, 6th months
  Transverse plane femoral cartilage thickness from three landmarks (from articular cartilage pothole,from midpoint of medial border and pothole of cartilage, from midpoint of lateral border and pothole of cartilage). Measured in millimeters. The sum of three points indicate a total thickness. A higher measurement indicates a thicker cartilage representing a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Teoman Aydın, Prof, MD, Study Director — Bezmialem Vakif University; Ozan Volkan Yurdakul, MD, Principal Investigator — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakif University, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cole BJ, Karas V, Hussey K, Pilz K, Fortier LA. Hyaluronic Acid Versus Platelet-Rich Plasma: A Prospective, Double-Blind Randomized Controlled Trial Comparing Clinical Outcomes and Effects on Intra-articular Biology for the Treatment of Knee Osteoarthritis. Am J Sports Med. 2017 Feb;45(2):339-346. doi: 10.1177/0363546516665809. Epub 2016 Oct 21. PMID 28146403
- [Background] Keen HI, Hensor EM, Wakefield RJ, Mease PJ, Bingham CO 3rd, Conaghan PG. Ultrasound assessment of response to intra-articular therapy in osteoarthritis of the knee. Rheumatology (Oxford). 2015 Aug;54(8):1385-91. doi: 10.1093/rheumatology/keu529. Epub 2015 Feb 16. PMID 25691769